CLINICAL TRIAL: NCT00244062
Title: "Brief Alcohol Intervention: The Healthy Moms Project."
Brief Title: Healthy Moms Alcohol Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 5R01AA012522-03 (NIH); 5R01AA012522-03 (NIH)
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2011-04

CONDITIONS: Fetal Alcohol Syndrome; Pregnancy; Alcoholism
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Alcoholism | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: counseling

SUMMARY:
The study proposes to test the efficacy of a primary care-based brief intervention with women who resumed heavy drinking during the post-partum period and who used alcohol during a previous pregnancy. The trial will also examine the effects of tobacco use, illicit drug use, depression and domestic violence on alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing age (18-40) who drank alcohol during their previous pregnancy and who report drinking above recommended limits in the post partum period.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2001-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The aim is to conduct a randomized test of the efficacy of brief physician/nurse advice in reducing alcohol use, alcohol-related harm, and fetal alcohol exposure in subsequent pregnancies in a sample of high-risk post partum pts.

SECONDARY OUTCOMES:
To est. the prevalence of drinking in ethnic div. pop. post partum women who are pts in 60 practices in Dane, Waukesha, and Milwaukee counties;the effect of age, race, tobacco use, marital status, partner alcohol use, and readiness-to-change;

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fleming, MD, Principal Investigator — University of Wisconsin, Madison